CLINICAL TRIAL: NCT03397849
Title: Lifestyle Intervention Using Mobile Technology in Patients With High Cardiovascular Risk
Acronym: LIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Turkey (Other Government)
Collaborators: Turk Telekomunikasyon A.Ş., Istanbul, Turkey (Unknown)
Responsible Party: Principal Investigator, Ahmet İlker Tekkeşin, Principal investigator, Ministry of Health, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIGHT
Record Dates: First submitted 2017-12-07; First posted 2018-01-12 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Primary Prevention; Digital Health; Lifestyle Risk Reduction
Keywords: Primary prevention; Lifestyle intervention; Digital health; Cardiovascular disease prevention
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Patients that are randomized to usual care group will receive guideline-standardized medications and lifestyle recommendations. Cardiovascular risk management and compliance to medication and lifestyle recommendation will be assessed and controlled by three cardiologists in clinical visits performed at 6 and 12 months. For the necessary cases counseling to other specialities will be performed for smoke cessation and weight management.
  Each study patients that are randomized to IMT plus usual care group will receive a group of smart devices including mobile phone (Vestel Venus e2) (Vestel, Manisa, Turkey), wristband (Xiaomi band 2) (Beijing Xiaomi Technology Co., Beijing, China), weight scale (Bluecat, Yongkang Tiansheng Electronic Co., Zhejiang, China) and blood pressure monitor (Clever Chek TD-3250) (TaiDoc Technology Co., Taipei County, Taiwan).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention using mobile technology (IMT) plus usual care (Active Comparator): Each study patients that are randomized to IMT plus usual care group will receive a group of smart devices including mobile phone (Vestel Venus e2) (Vestel, Manisa, Turkey), wristband (Xiaomi band 2) (Beijing Xiaomi Technology Co., Beijing, China), weight scale (Bluecat, Yongkang Tiansheng Electronic Co., Zhejiang, China) and blood pressure monitor (Clever Chek TD-3250) (TaiDoc Technology Co., Taipei County, Taiwan).
  Interventions: Behavioral: Intervention using mobile technology
- Only usual care (No Intervention): Patients that are randomized to only usual care group will receive guideline-standardized medications and lifestyle recommendations. Cardiovascular risk management and compliance to medication and lifestyle recommendation will be assessed and controlled by three cardiologists in clinical visits performed at 6 and 12 months. For the necessary cases counseling to other specialities will be performed for smoke cessation and weight management.

INTERVENTIONS:
Behavioral: Intervention using mobile technology — Each study patients that are randomized to IMT plus usual care group will receive a group of smart devices including mobile phone (Vestel Venus e2) (Vestel, Manisa, Turkey), wristband (Xiaomi band 2) (Beijing Xiaomi Technology Co., Beijing, China), weight scale (Bluecat, Yongkang Tiansheng Electronic Co., Zhejiang, China) and blood pressure monitor (Clever Chek TD-3250) (TaiDoc Technology Co., Taipei County, Taiwan)
  Arms: intervention using mobile technology (IMT) plus usual care

SUMMARY:
In the present study, investigators aim to compare intervention using mobile technology (IMT) plus usual care with only usual care in patients with a high risk for cardiovascular diseases (CVD). Investigators hypothesize that IMT plus usual care reduces the CVD risk and improves the secondary outcomes in this population through 12 months of follow-up period. Patients presented to the outpatient clinics in a tertiary hospital (Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Research and Training Hospital, Istanbul, Turkey) who were considered to be eligible according to inclusion and exclusion criteria will be enrolled to the study. The eligibility criteria is; Patients between 20 to 79 years old who are in high risk for CVD (10 years ASCVD risk ≥ 7.5%). Patients with prior CVD events (myocardial infarction, percutaneous coronary intervention, coronary artery by-pass grafting operation, stroke and peripheral artery disease), pregnancy, communication problems, severe neuropsychiatric problems and chronic kidney disease are excluded from the study. In addition, patients that are unable to use smartphone phone are also excluded.

ELIGIBILITY:
Inclusion Criteria:

* Presence of high risk for cardiovascular diseases (ASCVD risk score > 7.5%).

Exclusion Criteria:

* Patients with prior cardiovascular events including myocardial infarction, percutaneous coronary intervention, coronary artery by-pass grafting operation, stroke and peripheral artery disease.
* Pregnancy
* Patients with communication problems or severe neuropsychiatric problems
* Patients with chronic kidney disease
* Patients who are considered for being unable to use smart phone

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Atherosclerotic cardiovascular disease (ASCVD) risk score of individual patients at 12 months that is adjusted to baseline ASCVD risk score. | 12 months
  Patients with ASCVD risk score of >7.5 % are considered to have a high risk for 10-year atherosclerotic cardiovascular diseases.

SECONDARY OUTCOMES:
Smoke abstinence | 12 months
  Cessation of smoking habits including non-nicotine and electronic cigarettes during past 4 weeks will be measured at 12 months
Improvement in high sensitive C reactive protein levels (hs-CRP) (mg/L) (hs-CRP value at 12 months that is adjusted to baseline value) | 12 months
Improvement in quality of life | 12 months
  Quality of life will be evaluated by filling World Health Organization Quality of Life questionnaire. Minimum score is 122.77 and maximum score is 387.69 with higher values are considered as better quality of life.
Peak oxygen consumption value at 12 months that is adjusted to baseline value | 12 months
  Peak VO2 will be evaluated by cardio-pulmonary exercise testing
Major adverse cardiovascular events | 12 months
  Occurrence of death, myocardial infarction, Stroke, cardiovascular hospitalization
Systolic and diastolic blood pressure values (mmHg) at 12 months that are adjusted to baseline values | 12 months
Body mass index (BMI) (kg/m^2) level at 12 months that is adjusted to baseline level | 12 months
HbA1c (%) level at 12 months that is adjusted to baseline level | 12 months
Plasma fasting lipid levels (total cholesterol, low density lipoprotein, high density lipoprotein and trigliserid) (mg/dL) at 12 months that are adjusted to baseline levels | 12 months
Carotis intima-media thickness (mm) value at 12 months that is adjusted to baseline value | 12 months
  Carotis intima-media thickness will be evaluated by ultrasonography (USG)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Siyami Ersek thoracic and cardiovascular surgery research and training hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555